CLINICAL TRIAL: NCT03729999
Title: Ultrasound to Verify Lung-isolation During Single-lung Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Alok Moharir, Clinical Assistant Professor of Anesthesiology, Nationwide Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB18-01036
Record Dates: First submitted 2018-10-24; First posted 2018-11-05 (Actual); Results first posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Thoracic Diseases
MeSH Terms: conditions — Thoracic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Ultrasonography (Experimental): Patients requiring single lung ventilation for a surgical procedure will have a bedside ultrasound to evaluate lung isolation.
  Interventions: Device: Portable, Point-of-Care Ultrasound

INTERVENTIONS:
Device: Portable, Point-of-Care Ultrasound — Portable ultrasonography done at the bedside.
  Other Names: SonoSite

SUMMARY:
The purpose of the current study is to prospectively evaluate the usefulness of thoracic ultrasonography in demonstrating effective lung isolation during single-lung ventilation (SLV) in the pediatric patient. The primary hypothesis is that ultrasonography will accurately verify lung separation during SLV, as compared to fiberoptic bronchoscope (FOB).

ELIGIBILITY:
Inclusion Criteria:

* Requiring single lung ventilation for thoracic surgery

Exclusion Criteria:

* None

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-11-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ultrasonography
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ultrasonography
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 40
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 4.9 [0.7 to 14.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 40
Region of Enrollment [Number; unit: participants]
  United States | 40
Weight (kg) [Median (Inter-Quartile Range); unit: kilograms] | 18.0 [8.0 to 56.4]
Height (cm) [Median (Inter-Quartile Range); unit: centimeters] | 106 [69.8 to 170]
ASA physical status [Count of Participants; unit: Participants] — A grading system that assigns a class from I to VI, with higher numbers indicating a greater risk of complications
  Participants
    ASA I | 1
    ASA II | 12
    ASA III | 25
    ASA IV | 2
Technique for one lung ventilation (OLV) [Count of Participants; unit: Participants]
  Double-lumen tube | 16
  Bronchial blocker | 5
  Bronchial intubation | 19

OUTCOME MEASURES:

1. Primary Outcome: The Accuracy of Using Ultrasound to Assess Lung Isolation by Visualizing Lung Movement or Lack Thereof of Both the Operative and Non-operative Lung Fields.
Description: Ultrasound will be used to look for lung sliding in the ventilated lung field and lack of lung sliding and presence of lung pulse on the operative/isolated lung field. The effectiveness of this modality will also be compared to the lung auscultation for assessing lung isolation, which along with FOB is the current accepted standards of care.
Time Frame: Within 5 minutes of intubation and single lung ventilation device placement
Measure: Number (95% Confidence Interval); unit: percent
Groups:
- Auscultation: Patients requiring single lung ventilation for a surgical procedure will have auscultation via stethoscope to evaluate lung isolation.
Arm/Group | Ultrasonography | Auscultation
Number analyzed (Participants) | 40 | 40
percent
  Sensitivity | 97 [83.4 to 99.9] | 65 [46.5 to 79.7]
  Specificity | 67 [12.5 to 98.2] | 100 [31.0 to 100]
  Accuracy | 95 [82.7 to 98.5] | 68 [51.5 to 80.4]
  Positive predictive value (PPV) | 97 [83.4 to 99.9] | 100 [81.5 to 100]
  Negative predictive value (NPV) | 67 [12.5 to 98.2] | 20 [5.3 to 48.6]

2. Primary Outcome: Time to Confirm Lung Isolation
Description: Compare the time required to confirm lung isolation using auscultation, fiberoptic bronchoscopy (FOB), and ultrasound.
Time Frame: Within 5 minutes of intubation and single lung ventilation device placement
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Ultrasonography
Number analyzed (Participants) | 40
seconds
  Total FOB time | 179 [91 to 241]
  Total auscultation time | 21 [10 to 32]
  Total ultrasound time | 67 [46 to 142]

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Ultrasonography
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-19): https://cdn.clinicaltrials.gov/large-docs/99/NCT03729999/Prot_SAP_000.pdf